CLINICAL TRIAL: NCT03880851
Title: Single-arm Phase (II) Study on MR-based Hypofractionated Adaptive Image-guided Radiation Therapy for Prostate Cancer
Brief Title: MR-based Hypofractionated Adaptive IGRT of Prostate Cancer (M-base HyPro 2.0)
Acronym: Mbase_HyPro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Arndt-Christian Mueller, Deputy Head of the Department of Radiation Oncology, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mbase HyPro 2.0
Record Dates: First submitted 2019-02-11; First posted 2019-03-19 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: hypofractionation; MR-based IGRT; Mbase HyPro
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase II, Intervention: Plan adaption in case of significant changes of organ at risk or target volumes measured in weekly MRIs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated image-guided radiotherapy (Other): Hypofractionated image-guided radiotherapy "IGRT" to a total dose of 60 Gy (20 fractions) is performed.
  Weekly MRI are used to estimate volume/deformation changes of OAR and target volume.
  Intervention: In case of a significant change of target volume or OARs (threshold based) the radiation treatment plan is adapted on individual MR-anatomy.
  Interventions: Radiation: Plan adaptation of Radiation Treatment in case of anatomical changes

INTERVENTIONS:
Radiation: Plan adaptation of Radiation Treatment in case of anatomical changes — Image guided radiotherapy is given to 60Gy in 20 fractions. Intervention: Radiation treatment plan adaption in case of volume changes of target volume or not meeting OAR constraints due to volume changes.

SUMMARY:
Single-centre single-armed, non-randomized interventional phase II-study of hypofractionated image-guided radiotherapy "IGRT" with weekly magnetic resonance imagings "MRI" for personalized adaptation of the treatment plan depending on individual MR-anatomy of prostate/organ at risks "OAR" during course of IGRT.

DETAILED DESCRIPTION:
IGRT-schedule: 20 fractions to a total dose of 60 Gy

Personalized adaption of treatment plan dependning on volume-/ and constraint-thresholds and evaluation of biomarkers (multiparametric MRI, blood, tissue, stool, urine).

Treatment at MR-Linac allowed

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven prostate cancer with indication for RT
* cT1b-cT3a cN0 cM0
* ECOG Performance score 0-2
* IPSS≤12 (before planning computed tomography i.e. reached after neoadjuvant androgen deprivation therapy or tamsulosin)
* age>18 years
* Informed consent

Exclusion Criteria:

* not fulfilled inclusion criteria
* contraindication against curative RT
* age<18 years
* previous pelvic radiotherapy or planned pelvic radiotherapy
* comorbidities interfering with image-guided radiotherapy
* contraindications against multiparametric MRI (like hio prosthesis, pacer, allergy against contrast media)
* prior transurethral resection, highly focussed ultrasound or other pre-treatment of prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with gastrointestinal "GI" and genitourinary "GU" toxicity of >/= G2 | 2 years
  Hypothesis: reduction of GI/GU-toxicity (CTC-criteria 4.0, RTOG) from 20% to 10% at 2 years, power 80%

SECONDARY OUTCOMES:
Number of participants completing at least 2 of 4 MRI-examinations during course of IGRT | 6 months
  Feasibility and tolerability of completing at least 2 of 4 MRIs during treatment
Rate of participants achieving local control | 2, 5, 10 years
  In case of PSA progress: No evidence of local recurrence detected by MRI
Rate of participants achieving regional control | 2, 5, 10 years
  In case of PSA progress: No evidence of regional recurrence detected by MRI
Rate of participants achieving Distant-metastasis-free survival "DMFS" | 2, 5, 10 years
  No evidence of distant metastases diagnosed by cross-sectional imaging including bone scan, MRI, CT and PET
Number of Participants with biochemical no evidence of disease "bNED" | 2, 5, 10 years
  biochemical no evidence of disease according to Phoenix definition: nadir + 2ng/ml
Time without secondary treatment "TWIST" | 2, 5, 10 years
  Time without secondary treatment calculated from start of IGRT
CTC-Proctitis | 2, 5, 10 years
  CTC 4.0
CTC-Incontinence | 2, 5, 10 years
  CTC 4.0
Progression-free survival "PFS" | 2, 5, 10 years
  progression-free survival is defined as any progression (biochemical or other recurrences) or death or initiation of secondary treatment, calculation from start of IGRT
Overall survival "OS" | 2, 5, 10 years
  Overall survival is calculated from start of IGRT

CONTACTS AND LOCATIONS:
Locations (1):
- Müller Arndt-Christian, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided